CLINICAL TRIAL: NCT02729077
Title: PERIOPERATIVE RISK FACTORS FOR POSTOPERATIVE RESPIRATORY COMPLICATIONS IN PATIENTS AT RISK FOR OBSTRUCTIVE SLEEP APNEA
Brief Title: Risk Factors for Post-Operative Respiratory Complications in Patients at Risk for OSA
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Jyoti Pandya, Principal Investigator, Ohio State University
Other Study IDs: 2015H0052
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Respiratory Complications
MeSH Terms: interventions — Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Increased risk for OSA: Vital signs including oxygen saturation, respiratory rate, ECG, arterial pressure, BIS, blood pressure, heart rate will be monitored and hypoxemia will be measured during anesthetic care, and oxygen saturation and respiratory rate will be measured for 48 hours after surgery with pulse oximetry. Patients in this arm will be especially evaluated for hypoxemia and other complications.
  Interventions: Device: Pulse Oximetry
- Not increased risk for OSA: Vital signs including oxygen saturation, respiratory rate, ECG, arterial pressure, BIS, blood pressure, heart rate will be monitored and hypoxemia will be measured during anesthetic care, and oxygen saturation and respiratory rate will be measured for 48 hours after surgery with pulse oximetry.
  Interventions: Device: Pulse Oximetry

INTERVENTIONS:
Device: Pulse Oximetry — Use of pulse oximetry device for 48 hours after surgery.

SUMMARY:
This study investigates the incidence of postoperative respiratory complications (PRCs) including: oxygen desaturation events, tracheal re-intubations within 48 hours of surgery, and failure to wean from ventilator within 48 hours of surgery - in patients with and without risk factors for OSA undergoing elective, non-cardiac surgery (NCS).

DETAILED DESCRIPTION:
324 subjects will be enrolled into one of two groups: increased or not increased risk for OSA, n=162 patients per group. Preoperative assessments of OSA status, Mallampati score (an assessment for mouth and throat morphology), STOP-BANG test (assessment for risk of OSA), and medical history will be used to determine patient group assignment. All subjects will receive standard general anesthesia and monitoring as a part of standard of care whether or not she/he will participate in the study, including ECG, arterial pressure, SpO2, BIS, Blood pressure (BP), heart rate (HR), and respiratory rate (RR), all of which will be continuously recorded and data will be saved for every three minutes during induction using standard monitors. Standard monitoring assessments in PACU will be used, and patients with increased perioperative risk for OSA will be closely monitored for hypoxemia and other complications. The Nellcor Pulse Oximetry Sensor will be applied in PACU and continuously monitor the patient's oxygen saturation and respiratory rate for the first 48 hours postoperatively. At the end of the 48 hours, the device will be removed, and the de-identified data will be transferred to a computer with analysis software and examined for patterns in respiratory distress in both patient groups. Data collected from the Nellcor Bedside Respiratory Patient Monitoring System on pulse and oxygen saturation, as well as data on clinically significant events, such as PRCs, acute respiratory failure, tracheal reintubation, hypoxemia, CHF, MI, A-fib, and delirium will be analyzed to understand the effects of OSA on postoperative recovery

ELIGIBILITY:
Inclusion Criteria:

* Male or female , 18 to 75 years of age
* ASA I, II or III
* Capable and willing to consent
* Participants literate in English language

Exclusion Criteria:

* ASA IV or V
* Patients with severe visual or auditory disorder
* Illiteracy
* Chronic Obstructive Pulmonary Disease
* Restrictive Lung Diseases
* Benzodiazepines use
* Patients who were undergoing surgical procedures involving the upper airway, including tonsillectomy, septoplasty, uvuloplasty, uvulopalatoplasty, uvulopharyngoplasty, or uvulopalatopharyngoplasty, as these procedures were most likely to have been indicated to cure the primary disease process (OSA)
* Cardiac surgeries
* Neurosurgeries (Brain)
* Any condition, which in the opinion of the investigator would make subject ineligible for participation in the study such as history of unstable cardiovascular, pulmonary, renal, hepatic, neurologic (seizures), hematologic or endocrine abnormality (hyperthyroidism, unstable Diabetes type I/II)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients at Ohio State University Wexner Medical Center, aged between 18-75 years, with an American Society of Anesthesiologists (ASA) physical status of I (normal healthy patient), II (patients with mild systemic disease; no functional limitation) or III (patient with severe systemic disease; definite functional impairment - with relatively stable disease, but requiring therapy) who are scheduled to undergo elective surgeries under sevoflurane general anesthesia as a standard of care.
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2016-07; Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative respiratory complications (PRCs) based on cumulative minutes per 24 hours of oxygen desaturation events ≤ 90% | 24 hours
  Identify respiratory complications such as hypoxemia, respiratory failure requiring assisted ventilation, and reintubation, every 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicoleta Stoicea, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No